CLINICAL TRIAL: NCT06931184
Title: Self-Sampling In Cervical Cancer Routine Screening (FALCON)
Brief Title: Self- Sampling in Cervical Cancer Routine Screening
Acronym: FALCON
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Karolina Louvanto, Professor of Obstetrics and Gynecology, Tampere University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R23093
Record Dates: First submitted 2025-02-21; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-Sample (Other): Cervical cancer screening taken with self-sampling kit to increase the coverage of screening.
  Interventions: Other: self-sampling

INTERVENTIONS:
Other: self-sampling — increase screening coverage by self-sampling

SUMMARY:
SELF-SAMPLING IN CERVICAL CANCER ROUTINE SCREENING (FALCON) -Study implements a self-sampling option for the non-attendees of the national cervical cancer screening program in the Wellbeing Services County of Pirkanmaa. HPV primary testing is currently preferred method for cervical cancer screening. The HPV-DNA self-sampling has been shown to have screening performance equal to that of provider-obtained samples. In 2024, those turning 30, 35, 40, 45, 50, 55, 60, or 65 had the opportunity to participate in the FALCON study if they do not respond to the first invitation to cervical cancer screening. From March 2025 also women living in Kanta-Häme, Central Finland, Päijät-Häme, and Ostrobothnia can take part to the study.

The main objective of the FALCON study is to increase the current coverage of the cervical cancer screening program in the Pirkanmaa, Kanta-Häme, Central Finland, Päijät-Häme, and Ostrobothnia region and assess how acceptable self-sampling is for women.

ELIGIBILITY:
Inclusion Criteria:

* Women that do not respond to the first national cervical cancer screening invitation in 2024 and 2025 and to whom the reminder letter is sent to.
* Birth cohorts of women who will turn in screening year: 30, 35, 40, 45, 50, 55, 60 or 65 years old.

Exclusion Criteria:

* Women who do not belong to the screening year 2024 or 2025 invitation birth cohorts.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — woman
Enrollment: 40000 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in screening participation in a screening year | From baseline to the end of screening year, an average of 1 year
  Increase the cervical cancer screening coverage in the Wellbeing Services County of Pirkanmaa and women living in Kanta-Häme, Central Finland, Päijät-Häme, and Ostrobothnia via offering self-sampling option to those non-attendees and evaluate the self-sampling preference options among women.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital and Tampere University, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Time Frame: Beginning 3 months after publication with no end date
Access Criteria: IPD that underlie the results reported in a publication, after de-identification, will be available for researchers who provide a methodologically sound proposal with achievable aims. Proposals should be directed via e-mail to the PI of the study (KL); data requestors will need to sign a data access agreement.